CLINICAL TRIAL: NCT05389033
Title: Effect of Probiotic Supplementation on Exercise Metabolism During Exercise in the Heat and Subsequent Effect on Gastrointestinal Disturbance and Gut Microbiome Composition
Brief Title: Probiotic Supplementation and Exercise Performance in the Heat
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool John Moores University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro Heat LJMU
Record Dates: First submitted 2022-05-16; First posted 2022-05-24 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Acute Exercise; Probiotics

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active probiotic (Experimental): Lactobacillus acidophilus (CUL60 and CUL21), Bifidobacterium bifidum (CUL20), Bifidobacterium animalis subs p. Lactis (CUL34), 25 billion CFU, (Proven Probiotics, United Kingdom)
  Interventions: Dietary Supplement: Probiotic bacteria
- Placebo (Placebo Comparator): Chicory Root Extract (Min 90% Fructo-oligosaccharides) - Providing:
  100mg FOS Microcrystalline Cellulose - 137.26 mg
  Interventions: Other: Placebo Capsule

INTERVENTIONS:
Dietary Supplement: Probiotic bacteria — 28 days daily supplementation with active probiotic
  Arms: Active probiotic
Other: Placebo Capsule — 28 days daily supplementation with placebo
  Arms: Placebo

SUMMARY:
Endurance athletes will be invited to participate in the following study. Subjects will visit the laboratory on three occasions, each time following an overnight fast. Briefly, following an initial assessment and familiarisation, participants will be required to complete an endurance bout of cycling exercise in hot environmental conditions before and after 4 weeks of supplementing with a probiotic or placebo. During the exercise bouts, breath samples will be collected for measurements of whole-body metabolism, blood samples will be collected to assess serum metabolites and markers of gastrointestinal (GI) damage, and subjective measures of effort and symptoms of GI thermal distress will be collected. Before and after each exercise bout, participants will be required to provide a faecal sample for analysis of the microbiome and GI inflammation

DETAILED DESCRIPTION:
Study design

Participants The study is open to well-trained endurance 18-50 years (n = 24). Participants will be invited to take part in a matched-pairs design supplement intervention study. Participants will be split into two groups (n = 12), one which will supplement with a probiotic, the other a placebo, for 4 weeks.

Initial assessment During the first visit, subjects will first be asked that the have read the participant information sheet, including that they fit the inclusion criteria. Participants will then be asked to complete the Readiness to Exercise Questionnaire to ensure there are no contraindications before they proceed to exercising, such as a musculoskeletal injury or any medical condition for which exercise would pose an above normal risk (e.g. heart condition). Subjects will complete an incremental cycling test to volitional exhaustion to assess VO2max and blood lactate profile. Briefly, section 1 will commence at 95W and each stage will increase by 30W every 3 min. The wattage will continue to increase until the blood lactate concentration increases beyond 4mmol·L-1. The blood LT will be defined as the second abrupt increase of blood lactate concentration around 4mmol·L-1 by means of a linear-regression break point analysis. In the last 30s of each stage, heart rate (Polar Electro, Finland) will be recorded and a capillary blood sample (fingertip) will be obtained for blood lactate concentration analysis by micro-assay (Lactate Pro LT-1710, ArkRay Inc., Kyoto, Japan). This initial stage will be followed by a 15 min recovery period. Section 2 of the test protocol will then commence at 3.33 w/kg-1 for 150 s and thereafter will be increased by 50 W for a further 150 s. Subsequently, increases of 25 W every 60 s will occur until volitional fatigue or a drop in cadence below 70 rev/min-1. VO2max will be determined as the highest 30 s VO2 consumption.

After completing the initial VO2max test to determine exercise intensity and resting for 30-60 minutes, subjects will complete a familiarisation session during which they will cycle at the prescribed power output for 90 minutes followed by the time to exhaustion trial. This session will be used to familiarise subjects to the procedures of using a rectal thermometer, heart rate monitor, fluid consumption during exercise, exercise capacity test, and the timings of these throughout the experimental trial. The session will also be used to assess, and if necessary, adjust the velocity to attain the required 90% lactate threshold (~70-80% VO2max intensity).

Experimental trials On the morning of the main experimental trials at ~08:00, participants will report to the laboratory in a fasted state. A baseline blood (6 mL) and breathe sample will be collected before participants are provided with a standardized high-CHO breakfast (CHO: 2 g.kg-1 BM; PRO: 0.4 g.kg-1 BM; Fat: 0.2 g.kg-1 BM; comprising cereal, milk, orange juice, and a cake bar. This is representative of an elite real-world cyclists 'Race-day" breakfast (see Table 3.3) (Heikura et al., 2019; Muros et al., 2019; Morton, unpublished observations; Sánchez-Muñoz et al., 2016). Blood samples (6 mL) will be taken 15,30, 60, 90, 120, min postprandially via an indwelling cannula. Subjects will then be fitted with a heart rate monitor (Polar Electro, Finland) and be asked to measure nude body mass (SECA, Hamburg, Germany) in private. It will be explained to the participant that they need to weigh themselves in only their underwear and they will be shown to a private room in order to do this.

Immediately following this, the 180 minute cycle will commence. Participants will complete a 180 minute, steady state cycle (90% lactate threshold), in the heat (32 °C, and 40% humidity). Oxygen consumption will be sampled every 30 min throughout the trial using a metabolic cart. This will required participants to breath into a mouth piece while wearing a nose clip. Ratings of perceived exertion (RPE) and heart rate will also be recorded every 30 minutes. Ratings of perceived GI discomfort will also be assessed during the exercise using a validated subjective scale. Participants will consume 200mL before commencing exercise and then every 15 minutes during the 180 min steady state cycling. Drinks will contain dextrose and fructose in a ratio of 2:1. The total carbohydrate ingestion rate will be 90g per hour. This amount is similar to that consumed by elite cyclists during Tour Stage racing (Morton, unpublished observations; Heikura et al., 2019).

Blood (6 mL) and breathe samples will be collected every 30 minutes in order to quantify exogenous carbohydrate absorption and oxidation. Blood samples will be drawn via an indwelling cannula and breath samples will be collected directly from the mixing chamber of the metabolic cart.

Immediately following the 180-min submaximal cycle, participants will undertake a cycling capacity test whereby they will cycle at 150% LT to volitional exhaustion. No music will be played, and no physiological measurements will be taken during the cycling capacity test. The only available information to the participants will be the fixed power output and cadence.

Before each of the experimental visits, participants will be provided with a standardised 24hr diet to provide 8 g.kg BM CHO. This will be provided from a mixture of food and drinks.

Supplementation Participants will then be randomly assigned to receive either a probiotic supplement, or visually identical placebo. Probiotics are live bacterial compounds that have been researched based upon their positive effects on human health, e.g. digestive and immune health. They are commonly found in many fermented foods such as yogurts and sourdough bread. These bacteria can be cultivated and taken in more concentrated forms, such as supplements. These can vary in terms of the number of different strains per product (usually between 1 - 10+ strains) and the number of live bacteria (products can range from millions to hundreds of billion colony forming units). The probiotics used in this study are a commercially available probiotic (Lactobacillus acidophilus (CUL60 and CUL21), Bifidobacterium bifidum (CUL20), Bifidobacterium animalis subs p. Lactis (CUL34), 25 billion CFU, Proven Probiotics), and come in a single pill form. Participants will be required to consume one pill daily and will be provided all supplements at the start of the study. Participants will be told verbally about the dosing, and instructions will be clearly stated on the label of the bottle. However, since these bacteria typically exist within the digestive system before supplementation, there is no risk of 'overdosing'. Likewise, there is no risk of harm to children, should they access the supplements.

Stool sample collection Following each experimental visit, samples will be collected from participants. Participants will be provided with commercial kits (Fe-Col® Faecal Sample Collection Kits, UK) and provided with instructions on how to use the kit and store the samples until they are able to transport them to research team. Participants will be asked to store the samples in a -20C freezer until they are able to bring the sample back to the laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Training/competing in exercise/sport for a minimum of 4 hours per week

Exclusion Criteria:

* Free from current illness
* No history of diabetes, high cholesterol, uncontrolled asthma or history of heart disease
* Free from current musculoskeletal injury
* No history of and free from GI related clinical conditions (IBS, Chron's Disease)
* Not currently taking NSAIDs/Antihistamines/Immunosuppressive drugs
* Without history of gastric ulcers or other gastric problems
* Free from habitual use of NSAIDs i.e. 2 x per week for previous 1 month
* Have no allergy or intolerance to standardised meal foods or be adherent to kosher diet

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-07-15 (Actual); Primary Completion 2023-04-10 (Estimated); Study Completion 2023-04-10 (Estimated)

PRIMARY OUTCOMES:
Change in Gastro-Intestinal Disturbance Following Probiotic Supplementation | 4 weeks
  Subjective assessment of GI discomfort experienced during cycling effort in the heat pre- and post- 4-week probiotic supplementation
Change in Exogenous Glucose-Fructose Oxidation Following Probiotic Supplementation | 4 weeks
  During exercise carbohydrate will be administered and the uptake and utilization of this will be measured via gas analysis of breath, tracer detection will be compared pre- and post- 4-week probiotic supplementation.

SECONDARY OUTCOMES:
Change in time to exhaustion after 180 mins cycling exercise in the heat following probiotic supplementation | 4 weeks
  Participants will cycle at a wattage on the bike that is high enough to induce fatigue, they will cycle at this wattage until failure (inability to keep the pedals turning/voluntary stoppage). This will be compared pre- and post- 4-week probiotic supplementation.
Change in circulatory metabolites during exercise following probiotic supplementation | 4 weeks
  Glucose will be measured during exercise, this will be compared pre- and post- 4-week probiotic supplementation.
Change in circulatory metabolites during exercise following probiotic supplementation | 4 weeks
  Lactate will be measured during exercise, this will be compared pre- and post- 4-week probiotic supplementation.
Change in circulatory metabolites during exercise following probiotic supplementation | 4 weeks
  Insulin will be measured during exercise, this will be compared pre- and post- 4-week probiotic supplementation.
Change in circulatory metabolites during exercise following probiotic supplementation | 4 weeks
  Non-esterified fatty acids will be measured during exercise, this will be compared pre- and post- 4-week probiotic supplementation.
Change in circulatory metabolites during exercise following probiotic supplementation | 4 weeks
  Glycerol will be measured during exercise, this will be compared pre- and post- 4-week probiotic supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Jamie N Pugh, PhD, Principal Investigator — Liverpool John Moores University
Locations (1):
- Liverpool John Moores University, Tom Reilly Building, Byrom Street Campus, Liverpool, Merseyside, United Kingdom